CLINICAL TRIAL: NCT00022477
Title: A Phase II Study Of Epothilone B Analog BMS-247550 (NSC 710428D) In Patients With Advanced Colorectal Carcinoma
Brief Title: BMS-247550 in Treating Patients With Recurrent or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11003B; UCCRC-11003B; NCI-3670
Record Dates: First submitted 2001-08-10; First posted 2003-08-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-247550 (Experimental): IV administration of BMS-247550 once every 21 days
  Interventions: Drug: BMS-247550

INTERVENTIONS:
Drug: BMS-247550
  Other Names: ixabepilone, Ixempra®

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BMS-247550 in treating patients who have recurrent or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in patients with locally recurrent or metastatic colorectal cancer treated with BMS-247550.
* Determine the toxicity of this drug in these patients.
* Determine the duration of response, median and overall survival, and time to progression in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive BMS-247550 IV over 3 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 weeks.

PROJECTED ACCRUAL: A total of 21-50 patients will be accrued for this study within 8-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic or locally recurrent adenocarcinoma of the colon or rectum that is not amenable to potentially curative surgical resection
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * The following are not considered measurable lesions:

    * Lesions seen on colonoscopic examination or barium study
    * Bone metastases
    * CNS lesions
    * Ascites
* Failed prior combination therapy comprising fluorouracil, leucovorin calcium, and irinotecan for metastatic disease
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* ALT/AST no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No grade 2 or greater peripheral neuropathy
* No history of allergic hypersensitivity reaction to compounds containing polyoxyethylated castor oil (Cremophor EL) (e.g., paclitaxel or compounds of similar chemical or biological composition to BMS-247550)
* No other currently active malignancy (less than 30% risk of relapse and completed prior therapy) except non-melanoma skin cancer or carcinoma in situ of the cervix
* No uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy
* No concurrent colony-stimulating factors during first course of therapy

Chemotherapy:

* See Disease Characteristics
* Prior adjuvant chemotherapy allowed
* At least 4 weeks since prior cytotoxic chemotherapy and recovered
* No more than 1 prior chemotherapy regimen for metastatic disease
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent anticancer hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent therapeutic radiotherapy

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior surgery

Other:

* At least 30 days since prior investigational agents
* At least 7 days since prior cimetidine
* No other concurrent anticancer investigational agents, commercial agents, or therapies
* No concurrent unconventional therapy, food, or vitamin supplement containing Hypericum perforatum (St. John's Wort)
* No concurrent cimetidine
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-09; Primary Completion 2002-10 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Response rate of BMS-247550 in colon cancer | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L. Kindler, MD, Study Chair — University of Chicago
Locations (15):
- United States (15):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - LaGrange Memorial Hospital, LaGrange, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York